CLINICAL TRIAL: NCT01594268
Title: A Prospective, Open-label Study to Assess Safety of Certican in Kidney Transplant Patients
Brief Title: A Prospective, Open Label Study of CERtican in KIdney Transplantation
Acronym: CERKI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRAD001AKR10
Record Dates: First submitted 2012-05-04; First posted 2012-05-09 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplant
Keywords: kidney transplant; Certican
MeSH Terms: interventions — Everolimus

ARMS (1):
- Kidney transplantation patient (Other): Kidney transplantation patient; single arm
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — A prospective, open-label study to assess safety of Certican in kidney transplant patients

SUMMARY:
A prospective, open label study of CERtican in KIdney transplantation

ELIGIBILITY:
Inclusion criteria: (Each patient must meet all of the following criteria.)

1. Males and females aged 20-65 years inclusive (in Korean age) who is scheduled to receive a primary kidney transplant.
2. Patients who received explanation of the study overview and signed on the informed consent form of this study.
3. de novo patients who are going to receive a kidney transplant from a deceased (cold ischemic time (CIT) < 36 hours), living unrelated or related donor

Exclusion criteria (Any patient who meets any of the following criteria will not be able to participate in the study.)

1. Multi-organ transplant recipients (e.g. simultaneous kidney-pancreas transplant) or patients who previously received an organ transplant other than a kidney transplant
2. Patients who are scheduled to receive a kidney transplant from a zero-antigen mismatched donor, bilateral kidney donor, a non-heart beating donor or a donor aged over 60 years
3. Patients who should avoid potential exposure to everolimus due to acute or chronic severe allergy treatment or patients who have hypersensitivity to everolimus and drugs of similar chemical classes (e.g. macrolides)
4. Class 1 PRA>30% by CDC-based assay or Class 1 PRA>50% by flow cytometry or EIA
5. Recipients of a kidney from a ABO-incompatible live-donor or T-cell cross matching-positive donor
6. Thrombocytopenia<75,000/mm3, absolute neutrophil count<1,500/mm3, and/or leukopenia<4,000/mm3
7. Severe hypercholesterolemia (350mg/dl) or hypertriglyceridemia (>500mg/dl) (However, patients with controlled hyperlipidemia are eligible for the study.)
8. Use of other investigational drugs for 30 days before enrollment in the study
9. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years before enrollment in the study, regardless of whether there is evidence of local recurrence or metastases
10. Pregnant or nursing women, and women of child-bearing potential who have a plan to be pregnant or do not consent to select an appropriate method of birth control (e.g. oral contraceptives, hormone implant, IUD, diaphragm barrier, condom, abstinence, etc.) (women of child-bearing potential means women less than 2 years post-menopausal or not having hysterectomy or surgical management, i.e. bilateral tubal ligation or bilateral oophorectomy)
11. Presence of surgery or medical condition (except for current transplant) which may change absorption, distribution, metabolism, and excretion of the investigational product at the investigator's discretion and/or severe diarrhea, active gastrointestinal disease or uncontrolled diabetes
12. Patients who are HIV-, HCV-, and HBV positive
13. Recipients of an organ from a donor who is HBsAg-, HCV-, and HIV-positive
14. Evidence of drug or alcohol abuse
15. Severe restrictive or obstructive pulmonary disease
16. Patients with severe liver disease (AST, ALT or total bilirubin>2.5 times ULN including abnormal liver function test)
17. Patients with severe systemic infection requiring continuous therapy which may influence the objectives of the study at the investigator's discretion
18. Patients in whom continuous treatment may lead to clinically serious infection at the investigator's discretion or patients with other severe surgery complications or problems with continuous wound treatment
19. Patients who have a genetic problem including galactose intolerance, lapp lactase deficiency, and glucose-galactose malabsorption

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events | 12 weeks
  frequency of serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Suwon